







Version 2 20-Feb-19

Centre:

PIN:

**REC Number:** 

IRAS ID: 256260

## PARTICIPANT ASSENT FORM

This assent form is for young people aged 12-15

Please complete this form after you have read the Information Sheet or listened to an explanation about the research.

## Online PTSD treatment for Young People and their Carers (OPTYC): Case Series Dr Patrick Smith

| | Please initial b | initial box |
|---|---|---|
| 1. | I confirm that I have read the information sheet dated 13/12/18 (version 1.0) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | |
| 2. | I understand that my participation is voluntary. If I decide at any time during the research that I no longer wish to take part, I can tell the researchers and pull out and I don't have to give a reason. If I pull out it will not affect my medical care or legal rights. | |
| 3. | I understand that relevant data collected during the study may be looked at by individuals from King's College London, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | |
| 4. | I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. | |
| <ul><li>5.</li><li>6.</li></ul> | I understand that my relevant confidential information will be disclosed to appropriate professionals, including my GP, if a clinical or research worker on the study becomes concerned about my own, or someone else's safety. | |
| 7. | I agree to my General Practitioner being informed of my participation in the study and being involved in the study, including any necessary exchange of information about me between my GP and the research team. | |
| 8. | I understand that the information held and maintained by South London and Maudsley NHS Foundation Trust may be used to help contact me or provide information about my health status. | |









Version 2 20-Feb-19 Centre: PIN: REC Number: IRAS ID: 256260

9. I understand that because I am under 16 years old, I can provide my informed assent to take part in this study, but my parent/carer will also need to provide formal consent for me to take part. I agree to take part in the above study.

Name of Participant Date Signature

Name of Person taking consent Date Signature